CLINICAL TRIAL: NCT02655367
Title: The Effect of Oat Processing on Gastric Emptying and Satiety Induced After Consuming Porridge
Acronym: Oatmet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Quadram Institute Bioscience (Other)
Collaborators: Clinical Research and Trials Unit (Norfolk & Norwich University Hospital, UK) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: IFR08/2014
Record Dates: First submitted 2016-01-12; First posted 2016-01-14 (Estimated); Last update posted 2016-09-02 (Estimated); Status verified 2016-01

CONDITIONS: Metabolic Syndrome
Keywords: MRI; oats; porridge; satiety; GI hormones; processing
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Milled followed by flaked oats (Experimental): Participant consumes test meal consisting of porridge made from milled oats on study day 1, followed by porridge made from flaked oats on study day 2
  Interventions: Other: Flaked oats; Other: Milled oats
- Flaked followed by milled oats (Experimental): Participant consumes test meal consisting of porridge made from flaked oats on study day 1, followed by porridge made from milled oats on study day 2
  Interventions: Other: Flaked oats; Other: Milled oats

INTERVENTIONS:
Other: Flaked oats — Test meal consisting of 264g porridge made with flaked oats
Other: Milled oats — Test meal consisting of 264g porridge made with milled oats

SUMMARY:
This crossover study is designed to compare the gastric layering and rates of emptying and by inference rates of digestion of two different porridge meals prepared from either finely milled or flaked oats. On each of two study days, a total of 9 MRI scans will be taken, I baseline and 8 post meal, to assess gastric layering and emptying over three hours. Blood samples will also be taken periodically over the same period in order to determine changes in concentrations of circulating glucose, insulin and key gastrointestinal hormones. Participants will also be asked to complete a questionnaire at predetermined times to assess feelings of satiation.

DETAILED DESCRIPTION:
Eight participants will be recruited onto the study via the Human Nutrition Unit (HNU) Volunteer Database, advertising fliers and social media. Potential participants will be invited to IFR for a talk about the study, followed by health screening if they wish to participate. Written, informed consent will be taken by a member of the research team prior to undertaking any study related procedures.

Each participant will undergo 2 study days (min.7 days apart) and they will eat 2 types of porridge in a random order. Allocation of the order of the porridge meals will be done before the participants are recruited onto the study, using an online randomizer. On one occasion participants will consume porridge made from milled oats and on the other occasion porridge made from flaked oats. Participants will undergo 9 MRI scans of the stomach over a 3h post ingestion period, and after each scan a 4 ml blood sample will be collected via an intravenous cannula. Feelings of satiety will be assessed using a short VAS questionnaire at 9 intervals during the study day.

Study day participants will not be able to eat any food after 10.00pm on the evening prior to each study day, but they will be allowed water until they go to bed. Participants will be asked to record what they have eaten on the evening prior to study day 1, and they will be asked to eat the same foods on the evening before the second study day. Participants must not consume any breakfast on the morning of the study day, but they can drink up until 7 am. The study day will start at 9 am at the Radiology Department at the Norfolk and Norwich University Hospital. After cannulation and blood sampling, initial baseline MRI scans and VAS questionnaires, the participants will eat the allocated porridge (264 g) and drink the water provided (175 ml). They will then undergo 8 more MRI scans, have blood taken 8 more times and complete 8 satiety questionnaires at specific time points.

After completion of all MRI scans, blood sampling and satiety questionnaires, participants will be provided with a 500 ml bottle of water and a packed lunch.

ELIGIBILITY:
Inclusion Criteria:

* Male (hormonal status of women would introduce more variation within small group)
* Age 20-55y (people older than the upper age limit for the study, may suffer from degeneration of the GI tract, which would compromise our study data).
* BMI 19-35 kg/m2
* Apparently healthy
* Normally eat lunch and breakfast
* Willing to eat porridge type meal
* Willing to be cannulated and have blood samples taken
* Be able provide written informed consent

Exclusion Criteria:

Potential participants will be excluded if:

* They are line managed or supervised by any members of the study team either at IFR or NNUHFT Radiology.
* They are a student with a dependency on any member of the NNUHFT/ IFR study team.
* They are related to or living with any member of the study team (NNUHFT or IFR).
* They have an intense dislike of/ intolerance / allergy to any of the constituents of the test meal.
* They are smokers or have smoked within the last year (smoking affects satiety/hunger); this also includes e-cigarettes.
* They have been diagnosed with any long term illness requiring active treatment e.g. diabetes, cancer, cardiovascular disease.
* They have had surgery on the stomach or intestine or suffered from oesophageal or gastrointestinal disease, whether diagnosed or self-reported.
* They currently suffer from, or have suffered from an eating disorder.
* They are taking antibiotics on a long-term basis.
* They regularly (more than once in 10 days) use antacids, laxatives.
* They have any problems with swallowing.
* They take prescribed or over the counter medication for digestive or gastrointestinal conditions.
* They are receiving anticoagulant therapy or have finished anticoagulant therapy within the previous week.
* They are taking any dietary supplements/ herbal remedies which may affect the study data unless they are willing to stop taking within the appropriate timescale for the study. These will be assessed on an individual basis.
* They are currently using Ginko supplements (unless the individual is willing to stop taking the supplements for a minimum of 1 week before screening and for the duration of the study).
* They are taking part in another research study (other than a questionnaire based study).
* Their blood pressure greater than 160/100 mmHg or less than 90/50 or 95/55 mmHg if symptomatic.
* They have any special dietary requirements (e.g. dairy-free).
* They have participated in a research study during the previous four months where the combined blood sampling from previous study and this study would exceed 470 ml.
* Any of the clinical screening results are indicative of a health problem which could affect the participants' well-being or which would affect the study data if they took part.
* The HbA1c result greater than 42 mmol/ ml.
* They are unwilling or unable to provide GP details.
* They refuse to give permission to inform GP of participation in study.
* They are not registered with a GP in the UK
* They have recently experienced unexplained weight gain or loss.
* They have a history of back problems or any other condition which limit ability to repeatedly sit up and lie down.
* They have a Hiatus Hernia.

MRI scanning specific exclusion criteria:

Potential participants will also be excluded from the study if they:

* Have a cardiac pacemaker or artificial heart valve.
* Have had any surgery in the last 6 months.
* Have aneurysm clips (metal clips from surgery).
* Have an implant, pump or any medical device in the body (e.g. cochlear implant, neurostimulator, intra-venticular shunt).
* Have worked with metals (using lathes or grinders) or sustained injury to eyes involving metal splinters or fillings.
* Have artificial eyes or limbs.
* Have been injured with shrapnel or bullets.
* Have a metal tattoo.
* Suffer from fits, blackouts or epilepsy.
* Suffer from claustrophobia.

Clinical screening exclusion criteria:

Potential participants will be excluded if clinical screening results deemed by the HNU Medical Advisor, to be indicative of a health problem which may compromise the well-being of the participant, or which could affect the study data.

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2015-11; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Volume of gastric content | 3 hours
  Three dimensional MRI data will be used to determine the volume of gastric content at each time point and thus allow the calculation of gastric emptying rate

SECONDARY OUTCOMES:
Satiety response | 3 hours
  A visual analogue scale questionnaire will be used to assess satiety response at each time point.

CONTACTS AND LOCATIONS:
Overall Officials: Alan R Mackie, PhD, Principal Investigator — Quadram Institute Bioscience
Locations (1):
- Institute of Food Research, Norwich, Norfolk, United Kingdom